CLINICAL TRIAL: NCT02892370
Title: An Open Label, Randomized, Two-period, Crossover Study to Assess the Effect of Food on SHR0302 and Mass Balance in Healthy Volunteers
Brief Title: Effect of a High-fat Meal on the Pharmacokinetics of SHR0302 and Mass Balance Study in Healthy Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SHR0302-103
Record Dates: First submitted 2016-09-02; First posted 2016-09-08 (Estimated); Last update posted 2016-09-08 (Estimated); Status verified 2016-09

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — ivarmacitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SHR0302 fasted to fed (Experimental): SHR0302 tablets (10 mg) administered on day 1 fasting, and day 7 with high fat, high calorie breakfast
  Interventions: Drug: SHR0302
- SHR0302 fed to fasted (Experimental): SHR0302 tablets (10 mg) administered on day 1 with high fat, high calorie breakfast, and day 7 fasting
  Interventions: Drug: SHR0302

INTERVENTIONS:
Drug: SHR0302 — SHR0302 tablets (10 mg)

SUMMARY:
The purpose of this open-label, randomized, two-period, two-treatment (single doses of 10 mg SHR0302 fasted or fed), crossover study was to evaluate the effect of a high-fat meal on the pharmacokinetics of SHR0302 and mass balance study in 14 healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male
* BMI:19-24 kg/m2, weight > 50 kg.
* Age:18-45

Exclusion Criteria:

* History of clinically significant laboratory results or disease.
* History of alcohol or drug abuse.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Estimated)
Dates: Start 2016-08; Primary Completion 2016-09 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
The maximum plasma concentration (Cmax) of SHR0302 | up to 72 hrs postdose
  up to 72 hrs postdose on day1 and day7
The area under the plasma concentration-time curve (AUC) of SHR0302 | up to 72 hrs postdose
  up to 72 hrs postdose on day1 and day7
The accumulative excretion rate of SHR0302 and its metabolites in urine and feces | up to 96 hrs postdose
  up to 96 hrs postdose on day1 and day7

SECONDARY OUTCOMES:
The number of volunteers with adverse events as a measure of safety | up to Day 21
  required last visit via telephone during D11 to D21

CONTACTS AND LOCATIONS:
Overall Officials: Chen Yu, BS, Principal Investigator — Shanghai Xuhui Central Hospital
Locations (1):
- Shanghai Xuhui Central Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided